CLINICAL TRIAL: NCT05810623
Title: Single-Dose Intravesical Instillation of Chemotherapy After Diagnostic/Therapeutic Flexible Ureteroscopy for Upper Tract Urothelial Carcinoma in the Prevention of Intravesical Recurrence: Prospective Randomized Multicenter Trial
Brief Title: Single-Dose Intravesical Chemotherapy After Diagnostic URS
Acronym: MINERVA
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: David D'Andrea (Other)
Responsible Party: Sponsor-Investigator, David D'Andrea, Priv. Doz. Dr., Medical University of Vienna
Organization: Medical University of Vienna (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2411-2021
Record Dates: First submitted 2023-03-31; First posted 2023-04-12 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-03

CONDITIONS: Upper Urinary Tract Urothelial Carcinoma; Bladder Cancer
Keywords: UTUC; intravesical chemotherapy; bladder cancer; recurrence
MeSH Terms: conditions — Urinary Bladder Neoplasms; Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- SI Chemotherapy (Experimental): Patients randomized to the experimental arm will receive a SI within 24h after diagnostic URS. In case of multiple diagnostic URS during the follow-up (including 2nd look for incomplete ablation, non-diagnostic first URS or UTUC recurrence) patients randomized to the interventional arm will receive a SI after each diagnostic URS for 2 years after the day of first diagnostic URS.
  Interventions: Drug: Intravesical Solution
- Observation (No Intervention): Patient randomized to the observational arm will be treated and followed according to institutional own standards.

INTERVENTIONS:
Drug: Intravesical Solution — Intravesical single dose instillation of chemotherapy within 24h from uretero-renoscopy
  Arms: SI Chemotherapy

SUMMARY:
Study design This study is a Phase III, randomized, open-label, multi-center, global study to determine the efficacy of a single immediate intravesical chemotherapy instillation (SI) in the prophylaxis of intravesical recurrence after diagnostic uretero-renoscopy (URS) of patients 18 years of age or older with the fist diagnosis of UTUC.

This study will randomize 394 patients globally Patients will be randomized in a 1:1 ratio to the interventional arm or to observation.

Study period This study will include a screening period, a treatment and disease assessment period, safety follow-up visits and a 5-year survival follow-up period to begin immediately after the treatment.

Screening period: The period up to 28 days prior to intervention during which the screening procedures occur.

Treatment and disease assessment period: The period starting the day of diagnostic URS (Day 0) during which patients receive their assigned treatment (Day 0 to day 1) and disease assessments are performed. All patients must follow the disease assessment schedule, which includes disease assessments at screening and every 3 months (±1 week) from the date of intervention until 24 months from the date of randomization, and then every 6 months for up to 5 years. The treatment and disease assessment period will end at the time of intravesical recurrence, death, or MINERVA-CTU decision to terminate the trial early.

Safety follow-up visits: Every patient in this study will be assessed for the occurrence of adverse events (AEs) and serious adverse events from the time of signed informed consent until 90 days after the administration of SI. All patients who receive SI will have safety visits 4, 8, and 12 weeks following administration of SI. Safety assessments include targeted physical examination, complications according to Dindo-Clavien classification and patient-reported outcomes (PRO) assessments.

Survival follow-up period: Patients will be followed up at in-clinic site visits, by telephone contact, or by contact with the patient's current physician for up to 5 years from the date of randomized into this study.

Objectives Primary objective Efficacy of a SI in the prophylaxis of intravesical recurrence after diagnostic URS for UTUC

Secondary objectives

* Time to intravesical recurrence
* 5-years intravesical recurrence rates
* Incidence of high-grade BCa recurrence
* Incidence and gravity of adverse events (AEs) due to the SI
* To collect and store blood, urine and tissue samples according to each country's local and ethical procedures for identifying candidate markers that may correlate with likelihood of clinical benefit (optional)
* To collect and store DNA according to each country's local and ethical procedures for future exploratory research into somatic mutations and genes/genetic variations that may influence oncologic outcomes, to study treatments and susceptibility to disease (optional)
* To assess disease-related symptoms and HRQoL in patients with UTUC treated with SI compared those undergoing observation
* To assess patient-reported treatment tolerability directly using specific PRO-CTCAE symptoms

Target study population The study population includes patients 18 years of age or older with a primary diagnosis of UTUC, scheduled for diagnostic URS

Duration of treatment Patients randomized to the interventional arm will receive a SI within 24h after diagnostic URS. In case of multiple diagnostic URS during the follow-up (including 2nd look for incomplete ablation, non-diagnostic first URS or UTUC recurrence) patients randomized to the interventional arm will receive a SI after each diagnostic URS for 2 years after the day of first diagnostic URS.

Follow-up of subjects post discontinuation of study treatment Patients who have discontinued study treatment due to toxicity, symptomatic deterioration, intravesical recurrence or investigator's decision will be followed up for survival until 5 years from the date of diagnostic URS.

Survival All randomized patients, regardless of disease status, will be followed up for survival until 5 years from the date of diagnostic URS.

Investigational product, dosage, and mode of administration Patients randomized to the interventional arm will receive a SI. The chemotherapy will be at investigator's discretion and institutional availability.

The selected chemotherapy must be approved by the MINERVA-CTU in discussion with the local investigator.

Statistical methods This study will randomize 394 patients globally. Patients will be randomized 1:1 to SI or observation.

Randomization will be stratified by the following factors:

1. Center
2. EAU UTUC risk stratification

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all the following inclusion criteria to participate in this study:

* Age ≥ 18 years
* Diagnosis primary localized UTUC
* Imaging examinations show no distant metastasis
* Patients who agree to receive SI after URS for UTUC and will undergo the standard treatment, postoperative management, and follow-up in accordance with current guidelines

Exclusion Criteria:

* Any concurrent systemic therapy for any cancer
* Prior bladder cancer within 5 years
* Prior radical cystectomy
* Concomitant bladder cancer
* Bilateral UTUC
* Pregnancy
* Patient refused to participate
* Life expectancy of less than one year
* Solitary kidney

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 394 (Estimated)
Dates: Start 2023-06-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Efficacy of a SI in the prophylaxis of intravesical recurrence after URS for UTUC | 2 years
  Proportion of patients free of intravesical recurrence at 2-years

SECONDARY OUTCOMES:
Time to intravesical recurrence | 5 years
  Time to first occurrence of an bladder tumor after URS for UTUC
5-years intravesical recurrence rates | 5 years
  Proportion of patients free of intravesical recurrence at 5-years
Incidence of high-grade BCa recurrence | 5 years
  Proportion of patients HG with intravesical recurrence at 5 years
Incidence and gravity of adverse events (AEs) due to the SI | 2 months
  Proportion of patients experiencing an AE
Biobanking | 10 years
  To collect and store blood, urine and tissue samples according to each country's local and ethical procedures for identifying candidate markers that may correlate with likelihood of clinical benefit
Genetic mutation analysis | 3 years
  Prevalence of lynch syndrome
To assess disease-related symptoms and HRQoL in patients with UTUC treated with SI compared those undergoing observation | 2 years
To assess patient-reported treatment tolerability directly using specific PRO-CTCAE symptoms | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No
IPD will be shared with other researchers once the trial will be completed. Project proposals must be submitted to the international coordinator committee for review